CLINICAL TRIAL: NCT05162495
Title: A Single Center, Two Arms, Non-interventional, Breath Samples Collection Clinical Trial, for Development of the TERA Bio Station T101, Intended for SARS-CoV-2 Exhalation Products Detection.
Brief Title: Breath Samples Collection Clinical Trial, for Development of the TERA BioStation T101, Intended for CoV-19 Exhalation Products Detection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tera Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TERA-COV-02
Record Dates: First submitted 2021-12-12; First posted 2021-12-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The participant's breath sample is taken by blowing preferably three times into a disposable TeraTube. Thereafter, the tube is sealed, sterilized, and scanned by the BioSafety Station for analysis of its bio-chemical spectral signature. This will take place once during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Requiring a diagnostic or screening RT-PCR test for COVID-19.
  Interventions: Device: BioStation T101 and TeraTube
- Arm B (Experimental): Positive to COVID-19 in RT-PCR test performed up to 48 hours before screening.
  Interventions: Device: BioStation T101 and TeraTube

INTERVENTIONS:
Device: BioStation T101 and TeraTube — Rapid detection of the novel SARS-CoV-2 (COVID-19) virus in breath samples.

SUMMARY:
The Sponsor has developed a rapid screening tool intended to determine if the subject tested has COVID-19.

DETAILED DESCRIPTION:
According to recent scientific literature, the virus infection occurs mainly through the nasal cavity, and therefore, samples of nasal and pharyngeal fluids are expected to be high viral load samples.

The proposed clinical trial is to test the mentioned for potential dominant virus particles absorbance frequencies according to which, it will be possible to perform a statistical analysis of spectral data of infected subjects' samples compared to healthy ones and to examine whether a statistical significance between 'Infected' and 'Healthy' can be demonstrated in terms spectroscopic measurements.

Indication for Use: Rapid detection of the novel SARS-CoV-2 (COVID-19) virus in breath samples.

The study is aimed to collect data in order to assess whether a patient's COVID -19 status can be identified by a unique spectrophotometric pattern.

ELIGIBILITY:
Inclusion Criteria:

General:

1. Male or female subject aged 18 years and above
2. Subject is able and willing to provide informed consent
3. Subject is able to complete the breath test.

   Arm A:
4. Requiring a diagnostic or screening RT-PCR test for COVID-19.

   Arm B:
5. Positive to COVID-19 in RT-PCR test performed up to 48 hours before screening.

Exclusion Criteria:

1. Male of female subject under the age of 18.
2. Subject is unable to provide and informed consent, for any reason.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | The collection of an additional samples requiring COVID 19 diagnostic evaluation will take approximately 1 minute from initial collection of the sample
  Rate of positive and negative cases in collected breath samples using breath analyzer test compare to PCR results.